CLINICAL TRIAL: NCT04566913
Title: Clinical And Radiographic Evaluation Of The Use Of Pontic Shield Technique For Alveolar Ridge Preservation In The Esthetic Region . A Case Series
Brief Title: The Use Of Pontic Shield Technique For Alveolar Ridge Preservation . A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ramy Mohamed Salah ELdin Thabet, Postgraduate, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101292
Record Dates: First submitted 2020-09-06; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: To Assess Bucco-lingual Dimension of the Ridge While Using Pontic Shield Technique as a Treatment Modality for Ridge Preservation

STUDY DESIGN:
Intervention Model Description: Case Series study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients recruited from Cairo University (Experimental): After Cone beam CT assessment , The patient is assigned for nonsurgical periodontal phase then an impression is taken for stent formation to facilitate tissue thickness measurement .
  > After 2 weeks , the patient is assigned for surgical phase to extract the palatal and apical aspect of the tooth and leave the buccal portion .
  Socket preservation is attempted in the socket , using 'genbioss ' bone graft. Modified free gingival graft is done on the pontic site to cover the buccal root shield and the bone graft .
  Post operative instructions include :
  1. Analgesics (Prufen 400 mg ) three times for three days
  2. Antibiotic (Augmentin 1gm ) twice daily for one week The patient will be assured to contact the operator of any unexpected complications occured .
  Interventions: Procedure: Pontic Shield Technique

INTERVENTIONS:
Procedure: Pontic Shield Technique — • Together the apical and the palatal portions of the root in the esthetic region will be delivered and the buccal part is left for assessment of stability of bucco-palatal dimension of alveolar ridge

SUMMARY:
To assess bucco-lingual dimension of the ridge while using pontic shield technique as a treatment modality for ridge preservation

DETAILED DESCRIPTION:
• Patients with non-restorable teeth in the esthetic area will be recruited from Faculty of Dentistry in Cairo University A pre-operative cone beam computed tomography ( CBCT ) will be taken to examine the non-restorable tooth , measure bucco-lingual width and exclude any fenestration or dehiscence in the labial bone plate

A non-surgical phase one therapy will be done for the patient as a preparatory phase

Proper oral hygiene measures and chlorohexidene mouthwash will be prescribed after the the first

Reassessment of the case to assure absence of any signs of inflammation and prescence of normal tissues before the surgical procedure

* The area will be anaesthetized using infiltration technique in labial site with 1.5ml of anaesthetic solution and palatal site with 0.3 ml of anaesthetic solution
* Decoronation of the tooth , if the crown is available, will be done to obtain a concave mesio-distal root
* A long shank root resection bur will be used to section the root mesiodistally as far apical as possible , in order to obtain the buccal half attached to the labial bone plate and together the apical and the palatal half will be attached to the palatal bone
* Periotome will be used to distort the periodontal ligaments between the palatal half of the root and palatal alveolar socket wall
* Together the apical and the palatal portions of the root will be delivered , using micro forceps
* Bone curettage will be done in the presence of peraipical infection
* Explorer will be used to exclude mobility of the buccal portion of the root
* The thickness of the buccal portion will be reduced to 2mm
* A large round bur will be used to reduce the height of the buccal portion in a mesiodistal direction.
* A bone grafting material will be placed in the remaining socket

ELIGIBILITY:
1-Inclusion Criteria:

1a- non-restorable teeth in the anterior esthetic zone

1b-Teeth not indicated for immediate implant placement for reasons such as acute periapical infection, insufficient buccolingual width, poor economical status

1c- Full mouth plaque score (FMPS )<25% at baseline

1d- Full mouth bleeding score (FMBS )<25% at baseline

1e -Systemically healthy

2-Exclusion Criteria:

2a- Fenestration or dehiscence in buccal plate 2b- Periodontally compromised tooth 2c- Mobility of the tooth or remaining root 2d- Smokers 2e- Pregnancy and lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Bucco-lingual ridge dimension | 6 months
  To assess the stability of the ridge after surgical procedure using bone calliper and CBCT via subtractive method technique

SECONDARY OUTCOMES:
Labial bone thickness | 6 months
  To assess the stability of labial plate after surgical procedure using CBCT via subtractive method technique
Gingival thickness | 3 months
  assess the the thickness of labial tissue using endodontic spreader to identify a numerical value

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The exact procedure and results of all outcome after finishing the study